CLINICAL TRIAL: NCT04099550
Title: Effect of Real-time Continuous Glucose Monitoring System in Overweight or Obese Adults With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, JEONG MI KIM, Assistant Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PNUHEnMJMK1
Record Dates: First submitted 2019-09-10; First posted 2019-09-23 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Continuous Glucose Monitoring; Prediabetic State; Obesity
MeSH Terms: conditions — Prediabetic State; Obesity

STUDY DESIGN:
Intervention Model Description: participants were randomised to undertake a 12-week lifestyle intervention with either RT-CGM or SMBG
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMBG with lifestyle intervention (Active Comparator): All participants receive a 12-week lifestyle intervention (diet and exercise). The control group was monitored self-monitoring blood glucose (SMBG) at least 2 times a day for initial 1-week.
  Interventions: Other: SMBG
- RT-CGM with lifestyle intervention (Experimental): All participants receive a 12-week lifestyle intervention (diet and exercise). The intervention group was monitored initial 1-week with a RT-CGM.
  Interventions: Device: RT-CGM

INTERVENTIONS:
Device: RT-CGM — The group was monitored blood glucose initial 1-week with a RT-CGM.
  Arms: RT-CGM with lifestyle intervention
Other: SMBG — The group was monitored self-monitoring blood glucose (SMBG) at least 2 times a day for initial 1-week.
  Arms: SMBG with lifestyle intervention

SUMMARY:
In Korea, 5 million adults aged 30 years or older have diabetes. The development and expansion of Korea's economy and society, has led to dramatic chances in people's lifestyle and diet habits, and an increase in life expectancy. However, changes in lifestyle and diet habits related to the improvements of socioeconomic status may contribute to an increased diabetes burden in Korea. Therefore, it is important to prevent diabetes.

The purpose of this study was to evaluate the effects of real time-continuous glucose measurement (RT-CGM) system compared to only lifestyle modification group on blood glucose, lipid profile and diabetes prevention in prediabetic adults with overweight or obesity.

DETAILED DESCRIPTION:
Optimising patient adherence to prescribed lifestyle interventions to achieve improved blood glucose control remains a challenge. Combined use of real-time continuous glucose monitoring (RT-CGM) systems may promote improved glycaemic control.

Thirty adult with overweight or obesity and pre-diabetes are randomised to using either RT-CGM or self monitoring of blood glucose (SMBG) for 1 week with lifestyle intervention.

After 3 month, outcomes were glycemic control (HbA1c, fasting glucose), weight, and lipid profile assessed pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ BMI 23 kg/m2
* impaired fasting glucose (fasting glucose 100 to 125 mg/dL) or impaired glucose tolerance (2-h plasma glucose during oral glucose tolerance test (OGTT) 140 - 199 mg/dl) or HbA1c 5.7% to 6.4%

Exclusion Criteria:

* type 1 diabetes or type 2 diabetes or undergoing treatment for diabetes
* clinical history including malignancy
* fast history of cardiovascular disease (e.g. myocardial infarction, stroke), surgery, and trauma which may affect blood glucose within last 6 months
* taking medication (e.g. glucocorticoid, antipsychotics, anticholinergic drug etc.) which affect blood glucose
* acute infection within last 1 month
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
HbA1C change | Outcomes were assessed at baseline (week 0) and end of intervention (week 12)
  All participants receive lifestyle intervention at week 0, week 4, and week 8. The intervention group was monitored initial 1 weeks with a RT-CGM and th control group continued self-monitoring blood glucose (SMBG) at least 2 times a day for 1 week.
  HbA1c at baseline (week 0) and end of intervention (week 12).
Weight (Kg) change | baseline (week 0) and end of intervention (week 12)
  weight change (Kg) at baseline (week 0) and end of intervention (week 12)

SECONDARY OUTCOMES:
lipid profile | baseline (week 0) and end of intervention (week 12)
  both groups were assessed fasting lipid profile (total cholesterol, triglyceride and HDL-cholesterol) at baseline (week 0) and end of intervention (week 12)

CONTACTS AND LOCATIONS:
Overall Officials: JEONG MI KIM, M.D, Principal Investigator — Pusan National University Hospital
Locations (1):
- Jeong Mi Kim, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gehlaut RR, Dogbey GY, Schwartz FL, Marling CR, Shubrook JH. Hypoglycemia in Type 2 Diabetes--More Common Than You Think: A Continuous Glucose Monitoring Study. J Diabetes Sci Technol. 2015 Apr 27;9(5):999-1005. doi: 10.1177/1932296815581052. PMID 25917335
- [Background] Murphy HR, Rayman G, Lewis K, Kelly S, Johal B, Duffield K, Fowler D, Campbell PJ, Temple RC. Effectiveness of continuous glucose monitoring in pregnant women with diabetes: randomised clinical trial. BMJ. 2008 Sep 25;337:a1680. doi: 10.1136/bmj.a1680. PMID 18818254
- [Background] Tanenberg R, Bode B, Lane W, Levetan C, Mestman J, Harmel AP, Tobian J, Gross T, Mastrototaro J. Use of the Continuous Glucose Monitoring System to guide therapy in patients with insulin-treated diabetes: a randomized controlled trial. Mayo Clin Proc. 2004 Dec;79(12):1521-6. doi: 10.4065/79.12.1521. PMID 15595336
- [Background] Chase HP, Kim LM, Owen SL, MacKenzie TA, Klingensmith GJ, Murtfeldt R, Garg SK. Continuous subcutaneous glucose monitoring in children with type 1 diabetes. Pediatrics. 2001 Feb;107(2):222-6. doi: 10.1542/peds.107.2.222. PMID 11158450
- [Background] Boland E, Monsod T, Delucia M, Brandt CA, Fernando S, Tamborlane WV. Limitations of conventional methods of self-monitoring of blood glucose: lessons learned from 3 days of continuous glucose sensing in pediatric patients with type 1 diabetes. Diabetes Care. 2001 Nov;24(11):1858-62. doi: 10.2337/diacare.24.11.1858. PMID 11679447
- [Background] Salkind SJ, Huizenga R, Fonda SJ, Walker MS, Vigersky RA. Glycemic variability in nondiabetic morbidly obese persons: results of an observational study and review of the literature. J Diabetes Sci Technol. 2014 Sep;8(5):1042-7. doi: 10.1177/1932296814537039. Epub 2014 May 29. PMID 24876453
- [Background] Dagogo-Jack S, Egbuonu N, Edeoga C. Principles and practice of nonpharmacological interventions to reduce cardiometabolic risk. Med Princ Pract. 2010;19(3):167-75. doi: 10.1159/000285280. Epub 2010 Mar 29. PMID 20357497
- [Background] Hedayati SS, Elsayed EF, Reilly RF. Non-pharmacological aspects of blood pressure management: what are the data? Kidney Int. 2011 May;79(10):1061-70. doi: 10.1038/ki.2011.46. Epub 2011 Mar 9. PMID 21389976
- [Background] Lindstrom J, Peltonen M, Eriksson JG, Ilanne-Parikka P, Aunola S, Keinanen-Kiukaanniemi S, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study (DPS). Improved lifestyle and decreased diabetes risk over 13 years: long-term follow-up of the randomised Finnish Diabetes Prevention Study (DPS). Diabetologia. 2013 Feb;56(2):284-93. doi: 10.1007/s00125-012-2752-5. Epub 2012 Oct 24. PMID 23093136
- [Background] Marquez-Celedonio FG, Texon-Fernandez O, Chavez-Negrete A, Hernandez-Lopez S, Marin-Rendon S, Berlin-Lascurain S. [Clinical effect of lifestyle modification on cardiovascular risk in prehypertensives: PREHIPER I study]. Rev Esp Cardiol. 2009 Jan;62(1):86-90. Spanish. PMID 19150019
- [Background] Yoon U, Kwok LL, Magkidis A. Efficacy of lifestyle interventions in reducing diabetes incidence in patients with impaired glucose tolerance: a systematic review of randomized controlled trials. Metabolism. 2013 Feb;62(2):303-14. doi: 10.1016/j.metabol.2012.07.009. Epub 2012 Sep 7. PMID 22959500
- [Background] Rosenberg K. Prediabetes Increases Risk of Cardiovascular Disease. Am J Nurs. 2017 Jun;117(6):71. doi: 10.1097/01.NAJ.0000520262.18448.1c. No abstract available. PMID 28541998
- [Background] Mayer-Davis EJ, Lawrence JM, Dabelea D, Divers J, Isom S, Dolan L, Imperatore G, Linder B, Marcovina S, Pettitt DJ, Pihoker C, Saydah S, Wagenknecht L; SEARCH for Diabetes in Youth Study. Incidence Trends of Type 1 and Type 2 Diabetes among Youths, 2002-2012. N Engl J Med. 2017 Apr 13;376(15):1419-1429. doi: 10.1056/NEJMoa1610187. PMID 28402773